CLINICAL TRIAL: NCT04318288
Title: Comparison of Different Anthropometric Parameters in Relation to Cardiometabolic Risk Factors in a Cohort of Subjects With Overweight and Obesity
Brief Title: Comparison of Anthropometric Parameters and Cardiometabolic Risk Factors Among Subjects With Overweight and Obesity
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Gianluigi Giannelli, Clinical Professor, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: 2/2020
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The study was aimed at comparing four different anthropometric parameters to cardiometabolic risk factors in overweight and obese subjects (Body Mass Index (BMI)≥25)

DETAILED DESCRIPTION:
the present study was focused to compare the level of statistical association among four different anthropometric parameters, body mass index (BMI), waist circumference (WC), waist to height ratio (WHtR) and neck circumference (NC) and the cardiovascular (CV) risk factors most commonly evaluated in the clinical practice such as systolic and diastolic blood pressure, and fasting glucose, lipid (triglycerides, total, High-density lipoprotein (HDL) and Low-density lipoprotein (LDL) cholesterol), insulin, Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), uric acid, 25-hydroxyvitamin D (25(OH)D), c-reactive protein (CRP), white blood cells and platelet number in a population of 1214 apparently healthy subjects with overweight and obesity subjects

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI> 25 Kg/m2)

Exclusion Criteria:

* Any kind of drug
* Hypertension
* Endocrine diseases (diabetes mellitus, hypo or hyperthyroidism, hypopituitarism, etc.),
* Chronic inflammatory diseases
* Renal failure
* Liver failure
* Angina pectoris
* Myocardial infarction and heart failure
* Genetic heart diseases
* Thrombocytopenias

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who came to the Outpatient Clinic of Nutrition at the National Institute of Gastroenterology "S. de Bellis," Research Hospital, Castellana Grotte, Italy.
Sampling Method: Probability Sample
Enrollment: 1214 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Body mass index | baseline
  Body mass index (BMI) (expressed in kg/m^2)
waist circumference | baseline
  waist circumference (WC) (expressed in cm)
neck circumference | baseline
  neck circumference (NC) (expressed in cm)
waist to height ratio | baseline
  waist to height ratio (WHtR)

SECONDARY OUTCOMES:
Intima-media thickness | baseline
  Intima-media thickness (IMT) (expressed in mm)
Blood pressure | baseline
  blood pressure (BP) expressed in mmHg
Total Cholesterol | baseline
  Total Cholesterol (expressed in mg/dL) concentration in serum
Triglyceride | baseline
  Triglyceride (expressed in mg/dL) concentration in serum
fasting blood glucose | baseline
  fasting blood glucose (FBG) (expressed in mg/dL) concentration in serum
HDL Cholesterol | baseline
  HDL Cholesterol (expressed in mg/dL) concentration in serum
Insulin | baseline
  Insulin (expressed in mg/dL) concentration in serum
Homeostasis model assessment: insulin resistance | baseline
  Homeostasis model assessment: insulin resistance index (HOMA-IR)
LDL Cholesterol | baseline
  LDL Cholesterol (expressed in mg/dL) concentration in serum
Platelets | baseline
  Platelets (expressed in 10^3/µL) concentration in serum
white blood cells | baseline
  white blood cells (WBC) (expressed in 10^3/µL) concentration in serum
Vitamin D | baseline
  Vitamin D (expressed in ng/dL) concentration in serum
C-reactive Protein | baseline
  C-reactive Protein (CRP) (expressed in mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Gastroenterology IRCCS S. de Bellis, Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No